CLINICAL TRIAL: NCT02299505
Title: A Multi-center, Randomized Open Label Study to Assess the Systemic Exposure, Effiacy, and Safety of 450 mg Ceritinib Taken With a Low-fat Meal and 600 mg Ceritinib Taken With a Low-fat Meal as Compared With That of 750 mg Ceritinib Taken in the Fasted State in Adult Patients With ALK Rearranged (ALK-positive) Metastatic Non-small Cell Lung Cancer (NSCLC)
Brief Title: Pharmacokinetic and Safety Study of Lower Doses of Ceritinib Taken With a Low-fat Meal Versus 750 mg of Ceritinib in the Fasted State in Adult Patients With (ALK-positive) Metastatic Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLDK378A2112; 2014-004001-32 (EudraCT Number)
Record Dates: First submitted 2014-11-14; First posted 2014-11-24 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: LDK378; ceritinib; Alk+; Alk positive; NSCLC; lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — ceritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ceritinib 450 mg with a low-fat meal (Experimental): Oral ceritinib QD (21 days/ cycle) at a dose of 450 mg (3×150 mg/capsule) administered in the morning immediately (within 30 minutes)following a low-fat meal.
  Interventions: Drug: ceritinib
- ceritinib 600 mg with a low-fat meal (Experimental): Oral ceritinib QD (21 days/ cycle) at a dose of 600 mg (4×150 mg/capsule) administered in the morning immediately (within 30 minutes) following a low-fat meal.
  Interventions: Drug: ceritinib
- ceritinib 750 mg on an empty stomach (Active Comparator): Oral ceritinib QD (21 days/ cycle) at a dose of 750 mg (5×150 mg/capsule) administered in the morning on an empty stomach (i.e., fasted from food and drink except water)
  Interventions: Drug: ceritinib

INTERVENTIONS:
Drug: ceritinib — The investigational drug ceritinib was supplied to the Investigators as 150 mg capsules, for oral administration.
  Other Names: LDK378

SUMMARY:
A Phase I study to assess the systemic exposure, effiacy, and safety of 450 mg ceritinib taken with a low-fat meal and 600 mg ceritinib taken with a low-fat meal as compared with that of 750 mg ceritinib taken in the fasted state in adult patients with ALK rearranged (ALK-positive) metastatic non-small cell lung cancer (NSCLC)

DETAILED DESCRIPTION:
This was an open-label, randomized, multi-center, parallel design, Phase I study in which the systemic exposure, efficacy and safety of ceritinib administered at 450 mg or 600 mg with a low-fat meal vs 750 mg in the fasted state was assessed in subjects with ALK+ NSCLC following multiple oral daily dosing of ceritinib. Subjects were randomized in a 1:1:1 ratio to once daily doses of oral ceritinib (450 mg following a low-fat meal, 600 mg following a low-fat meal or ceritinib 750 mg administered on an empty stomach). Randomization was stratified by brain metastases at Screening (presence or absence) and by prior treatment (prior crizotinib use with ALK+ determined by Fluorescent in situ hybridization (FISH); crizotinib-naïve but could be previously treated with other systemic anti-cancer therapy with ALK+ determined by FISH, or treatment-naïve subjects with ALK+ by IHC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of stage IIIB (and is not a candidate for definitive multimodality therapy) or IV ALK-positive NSCLC.
* Patients may have received one prior treatment regimen with crizotinib (all other ALK inhibitors are excluded).
* Patients may have received prior chemotherapy, biologic therapy, or other investigational agents. ALK inhibitors other than crizotinib are excluded.
* Patient has a World Health Organization (WHO) performance status 0-2.

Exclusion Criteria:

* Prior treatment with an ALK inhibitor other than crizotinib.
* History of carcinomatous meningitis.
* Presence or history of a malignant disease other than an ALK-positive advanced tumor that has been diagnosed and/or required therapy within the past 3 years.
* Clinically significant, uncontrolled heart disease and/or recent cardiac event (within 6 months)
* Patient has history of interstitial lung disease or interstitial pneumonitis, including clinically significant radiation pneumonitis (i.e., affecting activities of daily living or requiring therapeutic intervention).
* Patient has other severe, acute, or chronic medical conditions
* Patient is currently receiving treatment with warfarin sodium (Coumadin®) or any other coumarin-derivative anticoagulants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2015-04-09 (Actual); Primary Completion 2016-06-16 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of ceritinib | Study Day 22
  Pharmacokinetics (PK) parameters, including but not limited to AUClast, AUC0-24h, Cmax, Tmax, Tlast, Racc, and CLss/F

SECONDARY OUTCOMES:
Safety profile | The primary analysis will be based on data from all patients, up to the time at which all randomized patients have completed at least 12 weeks of ceritinib treatment or have discontinued study treatment, whichever is earlier.
  Gastrointestinal (GI) Adverse Events (AEs), all Serious Advers Events (AEs), vital signs, electrocardiograms (ECGs) and laboratory abnormalities
Plasma concentration of ceritinib | Study Day 1
  PK parameters, including but not limited to AUClast, AUC0-24h, Cmax, Tmax, Tlast, Racc, and CLss/F
Objective response rate (ORR) | Tumor assessments every 6 weeks until cycle 9. At least every 12 weeks thereafter until progressive disease.
  Recist v1.1; Cycle = 21 days
Duration of response (DOR) | Tumor assessments every 6 weeks until cycle 9. At least every 12 weeks thereafter until progressive disease.
  Recist v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (68):
- United States (7):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Loma Linda University, Loma Linda, California
  - Goshen Center for Cancer Care IU Health - SC, Indianapolis, Indiana
  - Maryland Oncology Hematology, P.A. SC-2, Rockville, Maryland
  - Essex Oncology of North Jersey PA SC, Belleville, New Jersey
  - Greenville Health System SC, Greenville, South Carolina
  - Utah Cancer Specialists Dept.of Utah Cancer Spec. (3), Salt Lake City, Utah
- Australia (2):
  - Novartis Investigative Site, Grafton, Auckland
  - Novartis Investigative Site, Auckland
- Novartis Investigative Site, Vienna, Austria
- Novartis Investigative Site, Edegem, Belgium
- Brazil (6):
  - Novartis Investigative Site, Natal, Rio Grande do Norte
  - Novartis Investigative Site, Passo Fundo, Rio Grande do Sul
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Itajaí, Santa Catarina
  - Novartis Investigative Site, Barretos, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Novartis Investigative Site, Sofia, Bulgaria
- Canada (4):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
- Novartis Investigative Site, Montería, Colombia
- Novartis Investigative Site, Brno, Czechia
- Germany (4):
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Würzburg
- Greece (2):
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Athens
- India (5):
  - Novartis Investigative Site, Hyderabad, Andhra Pradesh
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, Kolkata, West Bengal
  - Novartis Investigative Site, Delhi
- Italy (10):
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Meldola, FC
  - Novartis Investigative Site, San Giovanni Rotondo, FG
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Aviano, PN
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Novara
- Novartis Investigative Site, El Achrafiyé, Lebanon, Lebanon
- Malaysia (2):
  - Novartis Investigative Site, Kuching, Sarawak
  - Novartis Investigative Site, Pulau Pinang
- Novartis Investigative Site, Nieuwegein, Netherlands
- Poland (3):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Konin
  - Novartis Investigative Site, Tarnobrzeg
- Novartis Investigative Site, Saint Petersburg, Russia
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Spain (4):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Donostia / San Sebastian, Basque Country
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Madrid
- Taiwan (3):
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- Thailand (3):
  - Novartis Investigative Site, Hat Yai, Changwat Songkhla
  - Novartis Investigative Site, Bangkok, THA
  - Novartis Investigative Site, Bangkok
- Novartis Investigative Site, Talas / Kayseri, Turkey (Türkiye)
- United Kingdom (2):
  - Novartis Investigative Site, Metropolitan Borough of Wirral, Merseyside
  - Novartis Investigative Site, Newcastle upon Tyne, Newcastle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CLDK378A2112 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17802